CLINICAL TRIAL: NCT05923658
Title: How Clinicians Manage Their Patients Who May Need Antithrombotic Care
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Anthony Tang (Other)
Responsible Party: Sponsor-Investigator, Anthony Tang, Professor and Scientific Director, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Other Study IDs: Antithrombotic Care at the CCC
Record Dates: First submitted 2023-06-14; First posted 2023-06-28 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Thrombosis
Keywords: Clinical Practice Guidelines
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to assess the knowledge and provide an opportunity for education to clinician attendees of the Canadian Cardiovascular Congress (CCC) meeting using a series of simulated patient case scenarios.

DETAILED DESCRIPTION:
Health conditions requiring antithrombotic therapy are highly prevalent in Canada, contributing substantially to healthcare costs and patient quality of life. For example, over 60,000 Canadians will experience a heart attack per year.1 Alarming statistics such as this warrant appropriate treatment approaches from clinicians who specialize in cardiovascular conditions. The CCC is a national conference during which individuals with an interest or expertise in cardiovascular health from across the country attend. Leveraging this unique opportunity by implementing a simple educational endeavour during the 2023 event can provide instrumental insights on the most appropriate treatments recommended from the latest clinical practice guidelines to a wide set of practitioners; this could, in turn, potentially improve patient health outcomes.

This endeavour will take place at a set date from October 25th to 29th, 2023. Attendees of the CCC who approach a booth set up by the lead investigator of this project will be presented with the study letter of information and consent form on a tablet (i.e., an iPad). After providing an electronic informed consent to participate, a series of patient case scenarios that require antithrombotic care and therapy will be shown. For each case scenario, the attendee (now, considered a study participant) will be asked to indicate the treatment approach that he/she would choose. And finally, after reviewing all case scenarios and selecting the best treatment approach to his/her knowledge, the participant will be asked to provide an email address (which could be an anonymized one) to send the most appropriate treatment approaches for each case scenario. This last step allows the participant an educational opportunity to learn what the best practice approach is based on the most up-to-date clinical practice guidelines. The approximate total duration of the study is one-hour in total.

ELIGIBILITY:
Inclusion Criteria:

* Any clinician (i.e., licensed medical doctor, nurse practitioner) attending the CCC's 2023 event from October 25th-29th, 2023 will be included in this endeavour so long as they have the ability to provide informed consent (i.e., can read, write, and understand the English language).

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: By convenience, there will be approximately 5,000 attendees at this conference and it is expected that no more than 50% will participate in this study. Therefore, the expected total number of participants is 2,500.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Adherence to Clinical Practice Guideline Recommendations | 1-Month.
  Open-ended recommendations provided by all participants on how they would treat each patient case in each scenario will be qualitatively coded as follows: 1) adhering to the recommendations provided in the guidelines, 2) partly adhering the recommendations provided in the guidelines, and 3) not adhering to the recommendations provided in the guidelines. For each participant, a total score will be computed across all case scenarios to determine adherence level to the latest Canadian clinical practice guideline recommendations.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Antiperovitch P, Liu I, Mokhtar AT, Tang A. Evaluating Large Language Models in Cardiovascular Antithrombotic Care: Performance, Accuracy, and Implications for Clinical Practice. Can J Cardiol. 2025 Aug;41(8):1584-1591. doi: 10.1016/j.cjca.2025.04.008. Epub 2025 Apr 15. PMID 40239865